CLINICAL TRIAL: NCT00403988
Title: A Clinical Phase II Study of Vinorelbine and Oxaliplatin (Vinox) With or Without Trastuzumab (Herceptin®) in Advanced Breast Carcinoma
Brief Title: Vinorelbine and Oxaliplatin (Vinox) With or Without Trastuzumab (Herceptin®) in Advanced Breast Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The results of a same study design have shown low response with important side effects. Accordingly & ethicly, the study has been stopped.
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9116
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Oxaliplatin; Vinorelbine

INTERVENTIONS:
Drug: Oxaliplatin
Drug: vinorelbine

SUMMARY:
Study Objective :

To assess the efficacy and the safety of the combination of Oxaliplatin, and Vinorelbine with or without Trastuzumab as a salvage regimen in patients with Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, histologically or cytologically proven breast cancer.
* At least one bi-dimensionally measurable lesion.
* Previous treatment with chemotherapy as first line for metastatic disease is mandatory especially with anthracyclines +/- the Taxanes.
* Treatment as adjuvant is allowed.
* World Health Organization-ECOG performance status 0-2.
* Adequate renal function (Creatinine <= 1.4 or Creatinine clearance >= 30 ml/min)
* Adequate hepatic function (Liver Function Tests not more than 3 times the normal values)
* Adequate bone marrow reserve is required (Neutrophils (PMN) >= 2000/mm2 and Platelets >= 100,000/mm2)
* Patient who will receive Herceptin should have an over-expression of HER2-neu.

Exclusion Criteria:

* Symptomatic peripheral neuropathy (National Cancer Institute common toxicity criteria grade more than one).
* Pregnant or breast-feeding.
* History of prior malignancies (with the exception of excised cervical carcinoma-in-situ or non-melanoma cell skin carcinoma).
* Receiving or had received, any treatment with experimental drugs.
* Had known brain or leptomeningeal involvement.
* Had a serious medical condition like congestive heart failure or an Ejection Fraction ≥ 40 %.
* The presence of bone as a sole site of metastasis.
* Radiation therapy to all areas of measurable disease less than four weeks before treatment.
* Creatinine two times above the normal range
* Hypercalcemia
* Evaluable but not a measurable disease as a sole site of metastasis: pleural effusion - Ascites - Pericardial effusion.
* Concomitant steroid intake for > 4 weeks
* Bilirubin two times above the normal range

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-06; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
overall response rate | During the Study Conduct
time to progression (TTP). | during the study conduct

SECONDARY OUTCOMES:
survival | During the study conduct
tolerance | During the study conduct
toxicity. | During the study conduct

CONTACTS AND LOCATIONS:
Locations (1):
- AmericanUBMC, Beirut, Lebanon